CLINICAL TRIAL: NCT05807477
Title: Determination of SpO2 and PR Accuracy Specifications at Rest / Accuracy of Pulse Oximeters With Profound Hypoxia NIHO 19/ Pulse Oximeter Accuracy Evaluation Protocol
Brief Title: Accuracy of Pulse Oximeters With Profound Hypoxia At Rest (NIHO19)
Status: Completed | Type: Observational
Sponsor: Nihon Kohden (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 72Ag_Vital-00014
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-11

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adult healthy subjects: Adult healthy subjects capable of undergoing controlled hypoxemia to the levels outlined in the desaturation profile in an at rest state
  Interventions: Device: Pulse Oximeter

INTERVENTIONS:
Device: Pulse Oximeter — OLV-4202 pulse oximeter (SW version: 01-15)

SUMMARY:
The aim of this study is to determine the accuracy of devices called pulse oximeters, which measure blood oxygen by shining light through fingers, ears or other skin, without requiring blood sampling. Study will be used with patients at rest.

DETAILED DESCRIPTION:
This study is intended to evaluate performance of a new design pulse oximeter (test device) manufactured by Nihon Kohden Corporation sufficiently to support performance claims for an FDA 510K submission or ISO technical file. Specifically, SpO2 and pulse rate accuracy will be assessed for a Nihon Kohden OLV-4202 pulse oximeter with adult patients under a controlled setting of varying levels of inhaled oxygen concentration levels for patients at rest.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female subjects who can give written informed consent
* Healthy subjects capable of undergoing controlled hypoxemia to the levels outlined in the desaturation profile below
* Meeting the demographic requirements

Exclusion Criteria:

* Age below 18 or over 50
* Pregnant women
* Significant arrhythmia
* Blood pressure above 150 systolic or 90 diastolic
* Carboxyhemoglobin levels over 3%
* Subjects whom the investigator consider ineligible for the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers. At least 10 subjects will be recruited to complete the study. Of these 3 will be dark pigmented (FItzpatrick Scale Type 4, 5 or 6). If the number of samples is less than the required 200 or if less than 3 of dark pigment subjects successfully complete the study, subjects will be added to include 3 of dark pigmented subjects and at least 200 data points.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2024-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bickler, MD, PhD, Principal Investigator — UCSF Hypoxia Research Laboratory
Locations (1):
- UCSF Hypoxia Research Laboratory, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Data to be used by Sponsor only

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adult Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adult Healthy Subjects
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 2
  Multiethnic | 1
  Caucasian | 5
  Asian | 3
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor Oxygen Saturation by Arms Calculation
Description: Accuracy will be determined by comparing the noninvasive blood oxygen saturation measurement of the pulse oximeter (SpO2i) to that obtained from a blood sample (SRi) and calculating the arithmetic root mean square (Arms) error value as follows:
  Arms = Square root (sum of n samples of ((SpO2i - SRi) squared) / n)
Time Frame: 30 seconds
Population: Qualified subjects
Measure: Number; unit: percentage of SpO2
Arm/Group | Adult Healthy Subjects
Number analyzed (Participants) | 12
percentage of SpO2 | 2.0

2. Secondary Outcome: Accuracy of Sensor Pulse Rate by Arms Calculation
Description: Accuracy will be determined by comparing the noninvasive pulse rate measurement of the pulse oximeter (PRi) to the heart rate obtained from an electrocardiography reference device (HRRi) and calculating the arithmetic root mean square (Arms) error value as follows:
  Arms = Square root (sum of n samples of ((PRi - HRRi) squared) / n)
Time Frame: 30 seconds
Population: Qualified subjects
Measure: Number; unit: percentage of SpO2
Arm/Group | Adult Healthy Subjects
Number analyzed (Participants) | 12
percentage of SpO2 | 2.0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Adult Healthy Subjects
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
The study was reviewed and approved by the University of California at San Francisco Committee on Human Research. The approval letter is on file at UCSF.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT05807477/Prot_SAP_001.pdf